CLINICAL TRIAL: NCT02389660
Title: European Comparative Effectiveness Research on Internet-based Depression Treatment in Poland [Europejskie Badania Porównawcze Nad Efektywnością Interwencji Internetowej Dla Osób z Depresją] (E-COMPARED)
Brief Title: European Comparative Effectiveness Research on Internet-based Depression Treatment in Poland
Acronym: E-COMPARED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Social Sciences and Humanities, Warsaw (Other)
Collaborators: VU University of Amsterdam (Other); Linkoeping University (Other Government); University of Erlangen-Nürnberg (Other); London School of Hygiene and Tropical Medicine (Other); GGZ inGeest (Other); Universitat Jaume I (Other); Leuphana Universität Lünenberg (Unknown); University of Limerick (Other); University of Bern (Other); University of Valencia (Other); Inesc Porto (Unknown); Institut National de la Santé Et de la Recherche Médicale, France (Other Government); European Commission (Other); Ministry of Science and Higher Education, Poland (Other Government)
Responsible Party: Principal Investigator, Roman Cieslak, Vice-Rector for Research, University of Social Sciences and Humanities, Warsaw
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: W73/7. PR/2014
Record Dates: First submitted 2015-02-18; First posted 2015-03-17 (Estimated); Last update posted 2018-06-29 (Actual); Status verified 2018-06

CONDITIONS: Depression
Keywords: Depression, Blended Cognitive Behavioural Therapy, Internet intervention
MeSH Terms: conditions — Depression | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Blended CBT (Experimental): Internet based blended depression treatment combines individual face-to-face cognitive behavioural therapy (CBT) with CBT delivered through an Internet based treatment platform with mobile phone components. The core components of the CBT treatment are: (1) psycho-education, (2) cognitive restructuring, (3) behavioural activation, and (4) relapse prevention. These will be delivered over 13 sessions (6 online and 7 face-to-face, session sequence - alternate, online platform - Moodbuster).
  Interventions: Behavioral: Blended Cognitive Behavioural Therapy (CBT)
- Treatment as usual (Active Comparator): Treatment as usual (TAU) will be defined as the routine care CBT that subjects receive when they are diagnosed with depression in the setting of recruitment. We will not interfere with treatment as usual but we will monitor carefully which health care services are utilized by usual care patients using patient records and through self-report (including TIC-P measurements).
  Interventions: Behavioral: Treatment as usual

INTERVENTIONS:
Behavioral: Blended Cognitive Behavioural Therapy (CBT)
  Arms: Blended CBT
Behavioral: Treatment as usual
  Arms: Treatment as usual

SUMMARY:
Effective, accessible, and affordable depression treatment is of high importance considering the large individual and economic burden of depression. There is ample support for the effectiveness of Internet-based Cognitive Behavioral Therapy (CBT) for depression which is considered a promising alternative to routine depression treatment strategies. Most evidence comes from randomized controlled trials, however, and not from research in routine practice.

The European Comparative Effectiveness Research on Internet-based Depression Treatment (E-COMPARED) in Poland aims to compare the clinical and cost-effectiveness of blended CBT for adults with major depressive disorder (MDD) with treatment as usual (TAU). The trial will be conducted in routine mental health care in Poland, and is a part of the bigger project funded by European Commission (Grant Agreement No: 603098). In this randomized controlled trial, a total of 150 patients with MDD will be assigned to one of two conditions: 1) blended CBT, 2) TAU. Respondents in both conditions will be followed until 12 months after baseline (measures will be taken at baseline, 3 months, 6 months and 12 months).

DETAILED DESCRIPTION:
Introduction

Good mental health is of high value from an individual, economic and social perspective. Depression is a serious threat to such a good mental health and highly prevalent worldwide. On a yearly basis about 7% of the European population (around 30 million people) suffer from a major depression (MDD) (Wittchen et al., 2011). If we take subclinical forms of depression into account the prevalence rises up to 15%.

Depression is not only highly prevalent; it is marked by disabling emotional and physical symptoms. It has a severe negative impact on mental wellbeing, quality of life and social and work-related functioning of those who suffer from it both on the short and longer term. This impact equals at least conditions such as diabetes mellitus, heart disease and arthritis (Sprangers et al., 2000). Depression is associated with increased morbidity, mortality, health care utilization and health care costs. The World Health Organisation has predicted that depression will be the foremost overall cause of disability by 2030 (Mathers, & Loncar, 2006).

Objective

The main objective of the planned research is to compare the clinical and cost-effectiveness of blended Cognitive Behavioural Therapy (CBT) for adults with major depressive disorder (MDD) with treatment as usual (TAU).

Study design

The study is a two-arm randomised controlled non-inferiority and cost-effectiveness trial. The trial will be conducted in routine mental health care in Poland, and is a part of the bigger project funded by European Commission (Grant Agreement No: 603098). A total of 150 patients with MDD will be assigned to one of two conditions: 1) blended CBT, 2) TAU. Respondents in both conditions will be followed until 12 months after baseline (measures will be taken at baseline, 3 months, 6 months and 12 months).

Study population

A total of 150 patients with MDD will be recruited from routine clinical practice in Poland and will receive either depression treatment as usual or blended CBT depression treatment.

Treatment fidelity

To ensure treatment fidelity it is required that: (1) a detailed treatment manual is available to guide therapists through the treatment, (2) regular meetings are organized between the therapists and the research team to prevent drift, (3) therapists will register the number of sessions, the frequency of the sessions, the main strategies used in each session and the duration of each contact.

Randomization

Randomization will be conducted by an independent researcher who is not involved in the trial. Randomisation will take place at an individual level, stratified by country, after the eligibility and baseline assessment. The independent researcher will create the allocation scheme with a computerised random number generator (Random Allocation Software). The allocation ratio will be 1:1. We will use block randomization with variable block sizes that vary between 8 and 14 allocations per block. Subjects will be randomized into two groups: Internet based blended depression treatment or treatment as usual. All investigators and clinicians will be unknown to the randomization scheme.

Sample size calculation

Sample size calculation is based on the non-inferiority design and calculated for the primary clinical outcome symptoms of depression. 150 patients in Poland will enable us to detect a clinically significant effect size of d=0.24 (Cuijpers et al., 2014).

Statistical Analysis

Multiple imputation will be used to impute missing cost and effect data. Intention-to-treat analyses (ITT) increase the risk of type I errors in non-inferiority (NI) trials and non-intention-to treat analyses are preferred over ITT analyses in NI designs. Therefore, the primary statistical analyses will be per protocol analyses meaning that only those patients that have completed the treatment will be included in the analyses. ITT analyses will be used in sensitivity analyses to increase confidence in the results obtained by including all participants in the analyses independent of whether they have completed the treatment or not. Blended depression treatment is considered no less effective than care-as-usual when the two-sided 95% confidence interval (the range of plausible differences between the two treatments) lies entirely above the standard mean difference of 0.20 which is the non-inferiority margin and the smallest clinically acceptable difference.

ELIGIBILITY:
Inclusion Criteria:

* Meet DSM-IV diagnostic criteria for MDD as confirmed by the telephone administered MINI International Neuropsychiatric Interview version 5.0 and a score a score of 5 or higher on the PHQ-9 screening questionnaire.

Exclusion Criteria:

* Current high risk for suicide according to the MINI Interview section C
* Serious psychiatric co-morbidity: substance dependence, bipolar affective disorder, psychotic illness, obsessive compulsive disorder, as established at the MINI interview
* Currently receiving psychological treatment for depression in primary or specialised mental health care
* Being unable to comprehend the spoken and written Polish
* Not having access to a PC and fast Internet connection (i.e. broadband or comparable).
* Not having a Smart phone that is compatible with the mobile component of the intervention that is offered or not willing to carry a Smartphone if one is provided with one by the research team for the study duration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Depression at 12 months | Baseline, 12 months
  Symptoms of depression will be assessed with the 9-item self-report The Patient Health Questionnaire (PHQ) (Kroenke et. al., 2001).

SECONDARY OUTCOMES:
Change from Baseline Symptoms of Depression at 12 months | Baseline, 12 months
  Symptoms of depression will be assessed with the 16-Item Quick Inventory of Depressive Symptomatology (QIDS) (Rush et al., 2003).
Change from Baseline Diagnosis of Depression at 12 months | Baseline, 12 months
  A diagnosis of depression will be assessed with the MINI International Neuropsychiatric Interview (M.I.N.I) version 5.0. The M.I.N.I. is a structured diagnostic interview based on the Diagnostic and Statistical Manual of Mental Disorders (DSM-IV) and on International Classification of Diseases (ICD-10) criteria. The interview compares well with Structural Clinical Interview for DSM-IV disorders (SCID) (Sheehan et al., 1998) and the Composite International Diagnostic Interview (CIDI) (Lecrubier et al., 1997; Sheehan et al., 1998).
Change from Baseline Health Service Uptake and Production Loss Due to Illness at 12 months | Baseline, 12 months
  Health service uptake and production loss due to illness will be measured with the Trimbos and iMTA Questionnaires on Costs Associated with Psychiatric Illness (TiC-P; Hakkaart-van Rooijen, van Straten, Donker, Tiemens, 2002).
Therapeutic Alliance | 3 months
  The therapeutic alliance between therapists and patient will be assessed with the short version of the Working Alliance Inventory (WAI-SF; Hatcher & Gillaspy, 2006).
Patient's Satisfaction with the Treatment | 3 months
  Patient's satisfaction with the treatment was assessed with Client Satisfaction Questionnaire (CSQ-8; Nguyen, Attkinson, & Stegner, 1983).
Satisfaction with the Platform | 3 months
  Satisfaction with the platform will be evaluated with the System usability scale (SUS; Brooke, 1996).
Alliance between the Patient and Technologies | 3 months
  We will assess the alliance between the patient and technologies with an adapted version of the WAI-SF, the Technology Alliance Inventory (TAI-SF).
Patients' Expectancy of Treatment | Baseline
  Patients' expectancy of treatment will be assessed with the credibility and expectancy questionnaire of Devilly and Borkovec (2000).
Change from Quality of Life at 12 months | Baseline, 12 months
  Quality of life will be assessed with the EQ-5D-5L (EuroQol; Van Agt, Essink-Bot, Krabbe, & Bonsel, 1994).

CONTACTS AND LOCATIONS:
Overall Officials: Roman Cieslak, PhD, Principal Investigator — University of Social Sciences and Humanities
Locations (1):
- University of Social Sciences and Humanities, Warsaw, Poland

REFERENCES:
- [Background] Wittchen HU, Jacobi F, Rehm J, Gustavsson A, Svensson M, Jonsson B, Olesen J, Allgulander C, Alonso J, Faravelli C, Fratiglioni L, Jennum P, Lieb R, Maercker A, van Os J, Preisig M, Salvador-Carulla L, Simon R, Steinhausen HC. The size and burden of mental disorders and other disorders of the brain in Europe 2010. Eur Neuropsychopharmacol. 2011 Sep;21(9):655-79. doi: 10.1016/j.euroneuro.2011.07.018. PMID 21896369
- [Background] Sprangers MA, de Regt EB, Andries F, van Agt HM, Bijl RV, de Boer JB, Foets M, Hoeymans N, Jacobs AE, Kempen GI, Miedema HS, Tijhuis MA, de Haes HC. Which chronic conditions are associated with better or poorer quality of life? J Clin Epidemiol. 2000 Sep;53(9):895-907. doi: 10.1016/s0895-4356(00)00204-3. PMID 11004416
- [Background] Mathers CD, Loncar D. Projections of global mortality and burden of disease from 2002 to 2030. PLoS Med. 2006 Nov;3(11):e442. doi: 10.1371/journal.pmed.0030442. PMID 17132052
- [Background] Cuijpers P, Turner EH, Koole SL, van Dijke A, Smit F. What is the threshold for a clinically relevant effect? The case of major depressive disorders. Depress Anxiety. 2014 May;31(5):374-8. doi: 10.1002/da.22249. Epub 2014 Feb 22. PMID 24677535
- [Background] Nguyen TD, Attkisson CC, Stegner BL. Assessment of patient satisfaction: development and refinement of a service evaluation questionnaire. Eval Program Plann. 1983;6(3-4):299-313. doi: 10.1016/0149-7189(83)90010-1. PMID 10267258
- [Background] Devilly GJ, Borkovec TD. Psychometric properties of the credibility/expectancy questionnaire. J Behav Ther Exp Psychiatry. 2000 Jun;31(2):73-86. doi: 10.1016/s0005-7916(00)00012-4. PMID 11132119
- [Background] Hatcher R, Gillaspy J. Development and validation of a revised short version of the working alliance inventory. Psychotherapy Research 16(1): 12-25, 2006.
- [Background] Rush AJ, Trivedi MH, Ibrahim HM, Carmody TJ, Arnow B, Klein DN, Markowitz JC, Ninan PT, Kornstein S, Manber R, Thase ME, Kocsis JH, Keller MB. The 16-Item Quick Inventory of Depressive Symptomatology (QIDS), clinician rating (QIDS-C), and self-report (QIDS-SR): a psychometric evaluation in patients with chronic major depression. Biol Psychiatry. 2003 Sep 1;54(5):573-83. doi: 10.1016/s0006-3223(02)01866-8. PMID 12946886
- [Background] Sheehan DV, Lecrubier Y, Sheehan KH, Amorim P, Janavs J, Weiller E, Hergueta T, Baker R, Dunbar GC. The Mini-International Neuropsychiatric Interview (M.I.N.I.): the development and validation of a structured diagnostic psychiatric interview for DSM-IV and ICD-10. J Clin Psychiatry. 1998;59 Suppl 20:22-33;quiz 34-57. PMID 9881538
- [Background] Lecrubier Y, Sheehan DV, Weiller E, Amorim P, Bonora I, Harnett Sheehan K, Dunbar GC. The Mini International Neuropsychiatric Interview (MINI). A short diagnostic structured interview: reliability and validity according to the CIDI. European Psychiatry, 12(5): 224-231, 1997.
- [Background] Hakkaart-van Rooijen L, van Straten A, Donker M, Tiemans B. Manual Trimbos/iMTA questionnaire for costs associated with psychiatric illness (TIC-P). Rotterdam: Institute for Medical Technology Assessment. 2002
- [Background] Brooke J. SUS-a quick and dirty usability scale. In Usability Eval Ind. Volume 189. Edited by Jordan PW, Thomas B, Weerdmeester BA, McClelland IL. London: Taylor & Francis Ltd; 1996:189-194.
- [Background] van Agt HM, Essink-Bot ML, Krabbe PF, Bonsel GJ. Test-retest reliability of health state valuations collected with the EuroQol questionnaire. Soc Sci Med. 1994 Dec;39(11):1537-44. doi: 10.1016/0277-9536(94)90005-1. PMID 7817218
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Derived] Doukani A, Quartagno M, Sera F, Free C, Kakuma R, Riper H, Kleiboer A, Cerga-Pashoja A, van Schaik A, Botella C, Berger T, Chevreul K, Matynia M, Krieger T, Hazo JB, Draisma S, Titzler I, Topooco N, Mathiasen K, Vernmark K, Urech A, Maj A, Andersson G, Berking M, Banos RM, Araya R. Comparison of the Working Alliance in Blended Cognitive Behavioral Therapy and Treatment as Usual for Depression in Europe: Secondary Data Analysis of the E-COMPARED Randomized Controlled Trial. J Med Internet Res. 2024 May 31;26:e47515. doi: 10.2196/47515. PMID 38819882
- [Derived] van Genugten CR, Schuurmans J, Hoogendoorn AW, Araya R, Andersson G, Banos R, Botella C, Cerga Pashoja A, Cieslak R, Ebert DD, Garcia-Palacios A, Hazo JB, Herrero R, Holtzmann J, Kemmeren L, Kleiboer A, Krieger T, Smoktunowicz E, Titzler I, Topooco N, Urech A, Smit JH, Riper H. Examining the Theoretical Framework of Behavioral Activation for Major Depressive Disorder: Smartphone-Based Ecological Momentary Assessment Study. JMIR Ment Health. 2021 Dec 6;8(12):e32007. doi: 10.2196/32007. PMID 34874888
- [Derived] Kleiboer A, Smit J, Bosmans J, Ruwaard J, Andersson G, Topooco N, Berger T, Krieger T, Botella C, Banos R, Chevreul K, Araya R, Cerga-Pashoja A, Cieslak R, Rogala A, Vis C, Draisma S, van Schaik A, Kemmeren L, Ebert D, Berking M, Funk B, Cuijpers P, Riper H. European COMPARative Effectiveness research on blended Depression treatment versus treatment-as-usual (E-COMPARED): study protocol for a randomized controlled, non-inferiority trial in eight European countries. Trials. 2016 Aug 3;17(1):387. doi: 10.1186/s13063-016-1511-1. PMID 27488181